CLINICAL TRIAL: NCT03735290
Title: A Randomized, Open-label, Multi-center, Phase 1b/2 Trial Evaluating the Safety and Efficacy of Intratumorally-administered Ilixadencel in Combination With Checkpoint Inhibitor (CPI) in Advanced Cancer Subjects Who Are Candidates for CPI Therapy
Brief Title: A Study to Evaluate the Safety and Effectiveness of ILIxadencel Administered Into Tumors in Combination With Checkpoint Inhibitor (CPI) in Patients With ADvanced Cancer
Acronym: ILIAD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision made not to move to Phase 2
Sponsor: Mendus (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM-202
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Non-small Cell Lung Cancer
Keywords: immunotherapy; ilixadencel; checkpoint inhibitor; allogeneic; somatic cell therapy; dendritic cell; intratumoral; in situ
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Single arm phase 1b. Randomized phase 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1b: Cohort 1, ilixadencel + pembrolizumab (Experimental): 3 x 10⁶ DCs (Dendritic Cells) of ilixadencel, 2x over 4 weeks (w). Pembrolizumab I.V. q3w
  Interventions: Biological: ilixadencel; Drug: Pembrolizumab
- Phase 1b: Cohort 2, ilixadencel + pembrolizumab (Experimental): 10 x 10⁶ DCs of ilixadencel, 2x over 4 weeks. Pembrolizumab I.V. q3w
  Interventions: Biological: ilixadencel; Drug: Pembrolizumab
- Phase 1b: Cohort 3, ilixadencel + pembrolizumab (Experimental): 10 x 10⁶ DCs of ilixadencel, 3x over 10 weeks. Pembrolizumab I.V. q3w
  Interventions: Biological: ilixadencel; Drug: Pembrolizumab
- Phase 1b: Cohort 4, ilixadencel + pembrolizumab (Experimental): Ilixadencel 3 times over 10 weeks: 1st dose 20 x 10⁶ DCs ilixadencel; 2nd dose 10 x 10⁶ DCs; 3rd dose 10 x 10⁶ DCs. Pembrolizumab I.V. q3w
  Interventions: Biological: ilixadencel; Drug: Pembrolizumab
- Phase 2 exp. cohorts HNSCC/NSCLC/Gastric/GEJ (Experimental): Subjects with HNSCC, NSCLC, gastric or gastroesophageal junction (GEJ) adenocarcinoma. ilixadencel administered intra-tumorally up to 3 times over 10 weeks; dose determined after Phase 1b. Pembrolizumab I.V. q3w according to currently approved doses and indications.
  Interventions: Biological: ilixadencel; Drug: Pembrolizumab
- Phase 2 comparator cohorts HNSCC/NSCLC/Gastric/GEJ (Active Comparator): Subjects with HNSCC, NSCLC, gastric/GEJ adenocarcinoma receiving active treatment with pembrolizumab I.V. q3w according to currently approved doses and indications.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Biological: ilixadencel — Intra-tumoral injection
  Arms: Phase 1b: Cohort 1, ilixadencel + pembrolizumab; Phase 1b: Cohort 2, ilixadencel + pembrolizumab; Phase 1b: Cohort 3, ilixadencel + pembrolizumab; Phase 1b: Cohort 4, ilixadencel + pembrolizumab; Phase 2 exp. cohorts HNSCC/NSCLC/Gastric/GEJ
Drug: Pembrolizumab — Administered intravenously over 30 minutes, every 3 weeks, at a dose of 200 mg

SUMMARY:
Patients in the Phase 1b part of the study will be treated with ilixadencel at an increasing dose and frequency, in combination with standard doses and schedules of checkpoint inhibitor (CPI) pembrolizumab. The Phase 1b study will determine the optimal dose and schedule of ilixadencel. Patients in the Phase 2 part of the study will be randomly assigned to receive either ilixadencel (at the dose determined in Phase 1b) combined with the CPI, or only the CPI.

Note: Recruitment to Phase 1b of the study has been completed.

DETAILED DESCRIPTION:
Despite improvements achieved with the use of CPIs, 50-80% of cancer patients do not respond to this therapy. There is growing evidence that combining CPIs with other forms of immunotherapy has the potential to improve the desired effects of both CPIs and immunotherapies. This study looks at the safety and effectiveness of the immunotherapy ilixadencel when used in combination with a CPI. A Dose-escalation Committee (DEC) will monitor the study for any significant safety issues during Phase 1b.

Note: Recruitment to Phase 1b of the study has been completed.

The study did not move forward to Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent.
* Must have histologically confirmed and specific (Human Papilloma Virus) HPV-positive or HPV-negative squamous cell carcinoma of the head and neck (SCCHN), non-small-cell lung cancer (NSCLC) or gastric or gastroesophageal junction (GEJ) adenocarcinoma. Patients with other tumor types who are candidates for pembrolizumab therapy (according to the FDA-approved prescribing information at the time of inclusion) can also be enrolled in Phase 1b. Tumor histology and most recent pathology report must be in subject's medical record. Tumor samples and/or biopsies will not be collected as part of this study.
* Eligible for pembrolizumab treatment per country-specific label and per physician's decision.
* ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1.
* Adequate organ function.
* Women of childbearing potential must follow contraceptive requirements; must have a negative pregnancy blood test at screening, and a negative blood or urine pregnancy test within 24 hours before each dose of ilixadencel; and must not be breastfeeding.
* Male subjects must agree to use condoms from screening until 90 days after the last dose of ilixadencel, or must have a female partner using a highly effective method of contraception as described above.

Exclusion Criteria:

* Prior history of invasive malignancy, unless complete remission has been achieved for at least 3 years and no additional therapy is required except for hormonal therapy or bisphosphonates.
* Active or previously untreated brain and/or leptomeningeal metastasis.
* Active autoimmune disease, pneumonitis or interstitial lung disease.
* Certain heart conditions including, but not limited to: Congestive heart failure; uncontrolled hypertension; unstable angina pectoris; pericarditis; myocarditis; mycardial infarction 6 months prior to study.
* Systemic immunosuppression except for replacement therapy.
* Life expectancy of less than 3 months.
* Any prior treatment with ilixadencel or prior treatment with anticancer agents (except pembrolizumab or other CPI for subjects in Phase 1b) within 4 weeks of starting study medication.
* Major surgery or significant traumatic injury within 4 weeks before study start.
* Known infection with human immunodeficiency virus (HIV).
* Active tuberculosis; active infection requiring anti-infective therapy (hepatitis with a negative viral load on maintenance will not be excluded).

Other protocol-defined inclusion/exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) (Phase 1b) | Up to Week 27
  Number of adverse events
Severity of adverse events (AEs) (Phase 1b) | Up to Week 27
  Grading per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Number of Dose Limiting Toxicities (DLTs) (Phase 1b) | Up to Week 27
  Dose Limiting Toxicities measured using CTCAE v5.0 and protocol DLT definition.
Number of subjects with clinically significant laboratory test abnormalities (Phase 1b) | Up to Week 27
  Grading per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Number of subjects with vital sign abnormalities (Phase 1b) | Up to Week 27
  Vital signs grading per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Antitumor Objective Response Rate (ORR) (Phase 2) | Up to Week 27
  Antitumor activity of ilixadencel plus CPI (checkpoint inhibitor) in each tumor type, centrally assessed using RECIST (Response Evaluation Criteria in Solid Tumors) v1.1

SECONDARY OUTCOMES:
Antitumor Objective Response Rate (ORR) RECIST 1.1 (Phase 1b and Phase 2) | Up to Week 27
  Antitumor activity of ilixadencel plus CPI (checkpoint inhibitor) in each tumor type, investigator and centrally assessed using RECIST (Response Evaluation Criteria in Solid Tumors) v1.1
Antitumor Objective Response Rate (ORR) iRECIST (Phase 1b and Phase 2) | Up to Week 27
  Antitumor activity of ilixadencel plus CPI (checkpoint inhibitor) in each tumor type, investigator assessed using iRECIST (Immune Response Evaluation Criteria in Solid Tumors)
Clinical Benefit Rate (Phase 1b and Phase 2) | Up to Week 27
  Rate of complete and partial response and stable disease by investigator and centrally assessed RECIST (Response Evaluation Criteria in Solid Tumors) v1.1
Duration of response (Phase 1b and Phase 2) | Up to 24 months after Cycle 1 Day 1
  Measured in weeks. Assessed using RECIST v1.1 and iRECIST
Time to Progression (TTP) (Phase 1b and Phase 2) | Up to 24 months after Cycle 1 Day 1
  Measured in weeks. Assessed using RECIST v1.1 and iRECIST
Progression-free Survival (PFS) (Phase 1b and Phase 2) | Up to 24 months after Cycle 1 Day 1
  Measured in weeks. Centrally assessed using RECIST v1.1
Overall Survival (OS) (Phase 1b and Phase 2) | Up to 5 years
  Measured in months
Frequency of adverse events (AEs) (Phase 2) | Up to Week 27
  Number of adverse events
Severity of adverse events (AEs) (Phase 2) | Up to Week 27
  Grading per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Number of Dose Limiting Toxicities (DLTs) (Phase 2) | Up to week 27
  Dose Limiting Toxicities measured using CTCAE v5.0 and protocol DLT definition.
Number of subjects with clinically significant laboratory test abnormalities (Phase 2) | Up to Week 27
  Grading per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Number of subjects with vital sign abnormalities (Phase 2) | Up to Week 27
  Vital signs grading per Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Petra Domeij, Study Director — Mendus
Locations (5):
- United States (5):
  - Site 1010, Coral Gables, Florida
  - Site 1006, Iowa City, Iowa
  - Site 1011, Louisville, Kentucky
  - Site 1004, Chapel Hill, North Carolina
  - Site 1009, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm